CLINICAL TRIAL: NCT01224405
Title: Androgen Deprivation Withdrawal Versus Maintenance and Intermittent Chemotherapy Versus Continuous in Prostate Cancer Patients With Castrate Resistant Disease
Brief Title: Prostate Cancer, Androgen Deprivation Withdrawal and Intermittent Chemotherapy
Acronym: PON-PC-02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento Scienze Cliniche e Biologiche Università di Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2010-019004-24
Record Dates: First submitted 2010-09-03; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-06

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment arm (Active Comparator): ten docetaxel cycles + maintenance androgen deprivation.
  Interventions: Drug: Docetaxel + LH-RH analogues
- suspension arm (Experimental): Ten Docetaxel cycles + stop androgen deprivation therapy
  Interventions: Drug: Docetaxel
- intermittent arm (Experimental): Intermittent Docetaxel
  Interventions: Drug: Docetaxel
- Continuous arm (Active Comparator): Continuous Docetaxel
  Interventions: Drug: Continuous Docetaxel

INTERVENTIONS:
Drug: Docetaxel + LH-RH analogues — Docetaxel will be administered at a dose of 75 mg/m2 per square meter as a 1-hour intravenous infusion on day 1 every 21 days in association to 5 mg of prednisone orally twice daily.
  In patients randomised to arms A up to 10 cycles of docetaxel will be planned in association to maintenance of LH-RH analogues administration.
  Arms: Treatment arm
Drug: Docetaxel — Docetaxel will be administered at a dose of 75 mg/m2 per square meter as a 1-hour intravenous infusion on day 1 every 21 days in association to 5 mg of prednisone orally twice daily.
  In patients randomised to arms B up to 10 cycles of docetaxel will be planned, in association to stopping LH-RH analogues.
  Arms: suspension arm
Drug: Docetaxel — Patients randomised in the arms AB1 (intermittent docetaxel) will suspend treatment after at least 4 cycles if their PSA level will be reduced >50%. Docetaxel treatment will be resumed when the serum PSA will rise by >50% from the lowest PSA level recorded and will be >10 ng/mL or when there will be other evidence of disease progression. PSA progression must to be confirmed with a second assessment after 2 weeks before deciding to resume docetaxel administration.
  Arms: intermittent arm
Drug: Continuous Docetaxel — Patients randomised in the arms AB2 (continuous docetaxel) will continue treatment up to ten cycles after even if their PSA level at 4 cycles will be reduced >50% or will reach a level <4 ng/mL.
  Arms: Continuous arm
Drug: Continuous Docetaxel — Patients randomised in the arms AB1(intermittent docetaxel) will continue treatment up to ten cycles even if their PSA level after 4 cycles will be reduced >50% or will reach a level <4 ng/mL.
  Arms: Continuous arm

SUMMARY:
The study includes the recruitment of patients with advanced prostate cancer resistant to chemical castration This is a multicenter prospective trial randomized phase III

DETAILED DESCRIPTION:
The study includes the recruitment of patients with advanced prostate cancer resistant to chemical castration This is a multicenter prospective trial randomized phase III This study design that includes a double randomizzzazione aims generally demonstrating non-inferiority in terms of survival of the suspension dell'ormonoterapia versus the maintenance and / or administration of intermittent versus continuous administration of chemotherapy in patients with prostate cancer resistant to chemical castration I started to line chemotherapy with Docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years,
2. histologically documented adenocarcinoma of the prostate,
3. written informed consent to the study,
4. Castrate resistant metastatic prostate cancer in the presence of castrate levels of testosterone (<50 ng/ml) and eligible to docetaxel chemotherapy. The condition of castrate resistant prostate cancer is the defined either as the documentation of a new metastasis or PSA increase more than 50% or increase more than 25% from a lower PSA value during previous hormone therapy in case of disease response or stabilization to previous hormone therapy, respectively. Absolute PSA increase should be greater than 5 ng/ml,
5. an elevated PSA level must have been documented within 4 weeks of initiating docetaxel chemotherapy,
6. more than 4 weeks since major surgery and fully recovered,
7. more than 4 weeks since any prior radiation with any toxicity attributable to radiation resolved to grade 1 or less,
8. more than 8 weeks since the last dose of strontium or samarium,
9. ECOG Performance Status more than/equal to 2,
10. life expectancy >6 months,
11. required initial laboratory values: absolute neutrophil count > 1500/ul Platelets > 100,000/ul., Hemoglobin > 8.0 g/dl, Creatinine, SGOT, SGPT less than 2.0 X upper limit of normal, Bilirubin less than/equal to upper limit of normal (ULN).
12. Appropriate patient compliance

Exclusion Criteria:

1. Patients with increased serum PSA levels with negative bone scan and CT scan.
2. Prior systemic chemotherapy for prostate cancer. Prior neoadjuvant or adjuvant chemotherapy is permitted if there was no evidence of disease relapse within 12 months of the last dose of chemotherapy,
3. Peripheral neuropathy >grade 1,
4. myocardial infarction or significant change in anginal pattern within the last 6 months, symptomatic congestive heart failure (NYHA Class III or higher) or uncontrolled cardiac arrhythmia,
5. patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80,
6. poorly controlled diabetes (fasting blood glucose >250) despite optimization of medical therapy, peptic ulcers or other contraindications to steroid therapy,
7. previous history of malignant disease with the exception of non melanoma skin cancer curatively treated,
8. significant neurologic or psychiatric diseases preventing patients to give a valid informed consent,
9. brain metastases,
10. prisoner status
11. because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded.

    -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
overall survival | six years
  The primary aim of the study will be the demonstration of non inferiority in terms of overall survival of stopping androgen deprivation therapy (arm B) versus maintenance androgen deprivation therapy (arms A) and intermittent docetaxel therapy (arm AB1) versus continuous docetaxel therapy (arms AB2) up to ten cycles.

SECONDARY OUTCOMES:
Toxicity | six years
  Toxicity graded according to NCI Criteria
Progression free survival | six years
  Progression free survival measured according to Prostate Cancer Clinical Trials Working Group
Quality of life | six years
  Quality of life evaluated according to FACT-P questionnaire
Pain | six years
  Pain response evaluated by Mc-Gill Pain Questionnaire
Cost Analysis | six years
  A cost minimization analysis will be performed in order to find if there is a treatment strategy that may achieve the same outcome for least cost. The analysis will focus on the direct medical costs of each treatment, collected at patient level.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, PHD, Study Chair — Medical Oncology - Hospital San Luigi Gonzaga Orbassano (TO) - Italy; Bruno Castagneto, MD, Study Director — Medical Oncology - Hospital San Giacomo of Novi Ligure (AL) Italy; Marcello Tucci, MD, Principal Investigator — Medical Oncology - Hospital San Luigi Gonzaga of Orbassano (TO) - Italy
Locations (32):
- Italy (32):
  - Davide Perroni, Saluzzo, Cuneo
  - Roberto Faggiuolo, Alba
  - Franco Testore, Asti
  - Mario Clerico, Biella
  - Andrea Martoni, Bologna
  - Massimo Aglietta, Candiolo (Torino)
  - Alberto Muzio, Casale Monferrato
  - Mario Botta, Casale Monferrato
  - Rodolfo Passalacqua, Cremona
  - Marco Merlano, Cuneo
  - Luigi Toniolo, Garbagnate Milanese
  - Sergio Bretti, Ivrea
  - Giovanni Ucci, Lodi
  - Pierfranco Conte, Modena
  - Carla Sculli, Mondovì
  - Oscar Alabiso, Novara
  - Bruno Castagneto, Novi Ligure
  - Giovanna Succu, Nuoro
  - Alfredo Berruti, Orbassano (Torino)
  - Luigi Dogliotti, Orbassano (Torino)
  - Luigi Cavanna, Piacenza
  - Giorgio Cruciani, Ravenna
  - Corrado Boni, Reggio Emilia
  - Riccardo Ratti, Sanremo
  - Francesco Ferrau, Taormina
  - Fausto Roila, Terni
  - Carlo Alberto Raucci, Torino
  - Guido Vietti Ramus, Torino
  - Libero Ciuffreda, Torino
  - Gianpiero Fasola, Udine
  - Sergio Cozzi, Verbania
  - Domenico Amoroso, Viareggio